CLINICAL TRIAL: NCT01532206
Title: Interleukin-10 Levels and Remote Ischemic Preconditioning in Acute Myocardial Infarction.
Brief Title: IL-10 Levels and Remote Ischemic Preconditioning in Acute Myocardial Infarction
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Steven P. Schulman, MD, Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00069912
Record Dates: First submitted 2012-02-09; First posted 2012-02-14 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Acute Myocardial Infarction
Keywords: Remote ischemic preconditioning; inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remote ischemic preconditioning (Experimental): Remote ischemic preconditioning performed with Blood pressure cuff insufflation
  Interventions: Other: Blood pressure cuff insufflation
- Standard of care (No Intervention): Standard of care

INTERVENTIONS:
Other: Blood pressure cuff insufflation — Blood pressure cuff will be inflated to a pressure of 200mmHg for 5 minutes. This will be repeated x 3, separated by 5 minutes.
  Arms: Remote ischemic preconditioning

SUMMARY:
Remote ischemic preconditioning has proven beneficial in patients undergoing percutaneous coronary intervention and coronary artery bypass surgery. Animal studies suggest remote ischemic preconditioning increases levels of interleukin 10. The investigators aim to determine whether remote ischemic preconditioning results in an increase in IL-10 levels in patients following acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

- Acute myocardial infarction

Exclusion Criteria:

- Cardiogenic shock Active ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-03; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Interleukin 10 levels | 24 hours following RIPC

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Schulman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States